CLINICAL TRIAL: NCT07069582
Title: Plasma and Breastmilk Exposures to Antituberculosis Drugs in Breastfeeding Women: an Open-label, Randomized, Six-arm, Single-dose, Pharmacokinetic Study
Brief Title: Pharmacokinetics of Antituberculosis Drugs in Breastfeeding Women
Acronym: PRiMe
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Faculty of Medicine Universitas Padjadjaran (Unknown)
Responsible Party: Principal Investigator, Dick Menzies, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIME_V.2.0
Record Dates: First submitted 2025-06-12; First posted 2025-07-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-07

CONDITIONS: Tuberculosis Infection; Healthy Volunteer; Breastfeeding
Keywords: Tuberculosis infection; Latent tuberculosis infection; TBI; LTBI; Breastfeeding women; Rifampicin; Levofloxacin; Rifapentine; Isoniazid; Bedaquiline
MeSH Terms: conditions — Latent Tuberculosis; Breast Feeding | interventions — Rifampin; Isoniazid; Levofloxacin; rifapentine; bedaquiline

STUDY DESIGN:
Intervention Model Description: Simple randomization will be performed, with a ratio of 1:1:1:1:1:1 for rifampicin at 10 mg/kg (RIF10), rifampicin at 20 mg/kg (RIF20), levofloxacin at 10-15 mg/kg (LFX10-15), rifapentine at 10 mg/kg (RPT10), isoniazid at 5 mg/kg (INH5), and bedaquiline at 40 mg (BDQ400).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 10 mg/kg rifampicin (RIF10) (Experimental): Single-dose rifampicin at 10 mg/kg body weight
  Interventions: Drug: Standard dose rifampicin
- 20 mg/kg rifampicin (RIF20) (Experimental): Single-dose rifampicin at 20 mg/kg body weight
  Interventions: Drug: High dose rifampicin
- 5 mg/kg isoniazid (INH5) (Experimental): Single-dose isoniazid at 5 mg/kg body weight
  Interventions: Drug: Standard dose isoniazid
- 10-15 mg/kg levofloxacin (LFX10-15) (Experimental): Single-dose levofloxacin at 10-15 mg/kg body weight
  Interventions: Drug: Standard dose levofloxacin
- 10 mg/kg rifapentine (RPT10) (Experimental): Single-dose rifapentine at 10 mg/kg body weight
  Interventions: Drug: Standard dose rifapentine
- 400 mg bedaquiline (BDQ400) (Experimental): Single-dose bedaquiline at 400 mg
  Interventions: Drug: Standard dose bedaquiline

INTERVENTIONS:
Drug: Standard dose rifampicin — Single-dose rifampicin at 10 mg/kg body weight
  Other Names: RIF10
  Arms: 10 mg/kg rifampicin (RIF10)
Drug: High dose rifampicin — Single-dose rifampicin at 20 mg/kg body weight
  Other Names: RIF20
  Arms: 20 mg/kg rifampicin (RIF20)
Drug: Standard dose isoniazid — Single-dose isoniazid at 5 mg/kg body weight
  Other Names: INH5
  Arms: 5 mg/kg isoniazid (INH5)
Drug: Standard dose levofloxacin — Single-dose levofloxacin at 10-15 mg/kg body weight
  Other Names: LFX10-15
  Arms: 10-15 mg/kg levofloxacin (LFX10-15)
Drug: Standard dose rifapentine — Single-dose rifapentine at 10 mg/kg body weight
  Other Names: RPT10
  Arms: 10 mg/kg rifapentine (RPT10)
Drug: Standard dose bedaquiline — Single-dose bedaquiline at 400 mg
  Other Names: BDQ400
  Arms: 400 mg bedaquiline (BDQ400)

SUMMARY:
This study is a sub-study of the SSTARLET trial (NCT06498414). The overall aim is to assess the pharmacokinetic profiles after taking a single dose of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline in breastfeeding women and the excretion of these drugs in breast milk, with the hope of including breastfeeding women in future clinical trials of TPT, including expanding the inclusion criteria of the SSTARLET trial. In this study, healthy breastfeeding women who fulfill the eligibility criteria will be enrolled from several primary health care centers in Bandung, which will be referred to the TB Research Clinic of the Universitas Padjadjaran, Bandung, Indonesia. Ten participants will be randomized to each of the following six study arms:

* Arm A: Single-dose rifampicin at 10 mg/kg body weight (RIF10).
* Arm B: Single-dose rifampicin at 20 mg/kg body weight (RIF20).
* Arm C: Single-dose isoniazid at 5 mg/kg body weight (INH5).
* Arm D: Single-dose levofloxacin at 10-15 mg/kg body weight (LFX10-15).
* Arm E: Single-dose rifapentine at 10 mg/kg body weight (RPT10).
* Arm F: Single-dose bedaquiline at 400 mg (BDQ400).

DETAILED DESCRIPTION:
Pregnant and breastfeeding women have been largely excluded from recent and ongoing clinical trials due to ethical concerns, limiting their access to the latest advancements in tuberculosis (TB) therapy. To support the development of short, effective tuberculosis preventive treatment (TPT) regimens lasting 1-2 months, a phase 2 adaptive clinical trial (SSTARLET trial) is being planned. This trial will evaluate three experimental regimens: two months of daily double-dose rifampicin; one month of daily levofloxacin and rifapentine; and either one month of daily isoniazid and rifapentine or a bedaquiline-containing regimen. The comparator will be the current standard of four months of daily rifampicin. The safest and shortest regimen will be selected for progression to a phase 3 trial. Inclusion of breastfeeding women in future trials of these regimens is intended; however, limited pharmacokinetic (PK) and safety data exist regarding the excretion of these drugs into breast milk, which is necessary to support their use in this population.

The current study aims to establish the PK profiles of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline in breastfeeding women and the excretion of these drugs in breast milk, with the hope of including breastfeeding women in future clinical trials of TPT. The specific objective of the study is to describe the PK profiles after a single dose of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline in plasma and breast milk of breastfeeding women.

In this study, healthy breastfeeding women who fulfill the eligibility criteria will be enrolled from several primary health care centers in Bandung, which will be referred to the TB Research Clinic of the Universitas Padjadjaran, Bandung, Indonesia.

The primary outcomes in this study are the total drug exposure, i.e., the area under the concentration-time curve from 0 to 24 hours after drug administration (AUC0-24) and peak concentration (Cmax) of single doses of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline in plasma and breastmilk of breastfeeding women, including the breast milk/plasma ratios for AUC0-24 and Cmax to estimate the external exposure of the drugs to breastfed infants. The secondary outcomes are PK measures of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline other than AUC0-24 and Cmax, including time to Cmax (Tmax), elimination rate constant (Ke), elimination half-life (t1/2), apparent clearance (CL/F), and apparent volume of distribution (Vd/F) in plasma and breast milk of breastfeeding women.

The study design is an open-label, randomized, six-arm, single-dose, intensive PK study, that will be performed at the TB Research Clinic of the Universitas Padjadjaran, Bandung, Indonesia. Six oral drug dosages will be evaluated: rifampicin 10 mg/kg (RIF10), rifampicin 20 mg/kg (RIF20), levofloxacin 10-15 mg/kg (LFX10-15), rifapentine 10 mg/kg (RPT10), isoniazid 5 mg/kg (INH5), and bedaquiline 400 mg (BDQ400). Simple randomization will be performed, with a ratio of 1:1:1:1:1:1 for RIF10, RIF20, LFX10-15, RPT10, INH5, and BDQ400. Venous blood and breastmilk samples will be collected for PK assessments of each of the study drugs. Ten participants will be assigned to each arm, with a total participants of 60.

ELIGIBILITY:
Inclusion Criteria:

Participants may enter the study if all of the following apply:

1. Healthy breastfeeding women aged 18 years or older, with a minimum of 3 months and a maximum of 24 months after delivery of a healthy baby, and are not currently diagnosed with either TB infection or TB disease.
2. Have a body weight between 25 and 100 kg.
3. Provide written informed consent.

Exclusion Criteria:

Participants may not enter the study if any of the following criteria apply:

1. Grade 3-4 abnormalities on baseline blood chemistry tests, including serum alanine aminotransferase (ALT), creatinine, or blood glucose.
2. Grade 3-4 abnormalities on baseline hematological tests, including white blood count, platelets, or hemoglobin.
3. Contraindications or history of hypersensitivity/intolerance to rifampicin, isoniazid, levofloxacin, rifapentine, or bedaquiline.
4. Taking concomitant medications for TB disease, TB infection, diabetes mellitus, hypertension, HIV, cardiac disease or any other chronic diseases.
5. Having a breastfed infant who was diagnosed with TB infection or TB disease and is currently on treatment.
6. Pregnancy
7. Have an active, acute illness at the time of study enrolment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breastfeeding women
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve from 0 to 24 hours (AUC0-24) | Day 1 following single-dose drug administration
  Total drug exposures in plasma and breast milk, i.e., the total area under the concentration-time curve from 0 to 24 hours (AUC0-24) after administration of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline.
Peak concentration (Cmax) | Day 1 following single-dose drug administration
  Peak concentration (Cmax) in plasma and breast milk after administration of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline.

SECONDARY OUTCOMES:
Time to Cmax (Tmax) | Day 1 following single-dose drug administration
  Time to Cmax (Tmax) in plasma and breast milk after administration of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline.
Apparent clearance (CL/F) | Day 1 following single-dose drug administration
  Apparent clearance (CL/F) in plasma and breast milk after administration of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline.
Apparent volume of distribution (Vd/F) | Day 1 following single-dose drug administration
  Apparent volume of distribution (Vd/F) in plasma and breast milk after administration of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline.
Half-life (t1/2) | Day 1 following single-dose drug administration
  Half-life (t1/2) in plasma and breast milk after administration of rifampicin, isoniazid, levofloxacin, rifapentine, and bedaquiline.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Menzies, MD, Principal Investigator — Research Institute of the McGill University Health Centre, Montreal, Canada
Locations (1):
- Universitas Padjadjaran, Klinik Penelitian Tuberculosis (TB Research Clinic), Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Protocol and consent form will be available for data sharing once approved by research ethical review board. A detailed plan for data sharing of other study documents and/or data is under definition and will be posted during the study.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol and consent form will be available once approval is received from the research ethical board and will remain available.
Access Criteria: Access criteria will be specified in the plan for data sharing, once available.